CLINICAL TRIAL: NCT06703346
Title: Evaluation of Safety and Antitumor Activity of Lete-Cel (GSK3377794) in HLA-A2+ Participants With NY-ESO-1 Positive Previously Treated Advanced (Metastatic or Unresectable) Synovial Sarcoma or Myxoid/Round Cell Liposarcoma
Brief Title: Study to Evaluate Safety and Antitumor Activity of Lete-Cel (GSK3377794) in HLA-A2+ Participants With NY-ESO-1 Positive Previously Treated Advanced (Metastatic or Unresectable) Synovial Sarcoma or Myxoid/Round Cell Liposarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 208467 Substudy 2
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-11

CONDITIONS: Neoplasms
Keywords: Adoptive T-cell therapy; Letetresgene autoleucel; Lete-cel
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Letetresgene autoleucel (Experimental)
  Interventions: Drug: Experimental: Letetresgene autoleucel

INTERVENTIONS:
Drug: Experimental: Letetresgene autoleucel — Drug: Letetresgene autoleucel Letetresgene autoleucel will be administered. Drug: Cyclophosphamide Cyclophosphamide will be used as a lymphodepleting chemotherapy. Drug: Fludarabine Fludarabine will be used as a lymphodepleting chemotherapy.

SUMMARY:
This trial will evaluate safety and efficacy of human engineered T-cell therapies, in participants with advanced tumors. This trial is a sub study of the Master study NCT03967223.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥10 years of age at the time of signing the informed consent.
* Participant scheduled to receive clinical drug product supply must also weigh ≥40 kg.
* Participant has a diagnosis of synovial sarcoma or myxoid/round cell liposarcoma, confirmed by local histopathology with evidence of disease-specific translocation.
* Participant has advanced (metastatic or unresectable) synovial sarcoma or myxoid/round cell liposarcoma. Unresectable refers to a tumor lesion in which clear surgical excision margins cannot be obtained without leading to significant functional compromise.
* Male or female. Contraception requirements will apply at the time of leukapharesis and treatment.
* Life expectancy ≥24 weeks
* Participant has confirmed evidence of a relevant disease-specific translocation per below:
* For synovial sarcoma, presence of a translocation involving chromosome 18 (SYT gene) and/or chromosome X (SSX1, SSX2 or SSX4 genes).
* For myxoid/round cell liposarcoma, presence of a translocation involving chromosome 12 (DDIT3 gene) and/or chromosome 16 (FUS gene) and/or chromosome 22 (EWSR1 gene).
* Participant is either currently being treated with or has completed at least one standard-of-care treatment including anthracycline-containing regimens (e.g., doxorubicin alone, doxorubicin with ifosfamide) for advanced (metastatic or inoperable) disease. Participants who are intolerant to anthracycline may receive ifosfamide alone unless intolerant to or ineligible to receive ifosfamide. Participants who received anthracycline-based therapy in the neoadjuvant/adjuvant setting and progressed will be eligible.
* Participant must be positive for HLA-A*02:01, HLA-A*02:05, and/or HLA-A*02:06 alleles by a validated test in a designated central lab prior to leukapheresis
* Participant's tumor has been pathologically reviewed by a designated central laboratory with confirmed positive NY-ESO-1 expression defined as ≥30% of cells that are 2+ or 3+ by immunohistochemistry.
* Left ventricular ejection fraction ≥45% with no evidence of clinically significant pericardial effusion.
* Performance status: for participants <16 years of age, Lansky >60, or for participants ≥16 and <18 years of age, Karnofsky >60, or for participants ≥18 years of age, Eastern Cooperative Oncology Group (ECOG) of 0-1.
* Participant must have adequate organ function and blood cell counts, within 7 days prior to the day of the leukapheresis procedure
* Participant is fit for leukapheresis and has adequate venous access for the cell collection
* Female participants of childbearing potential (FCBP) must have a negative urine or serum pregnancy test.
* Participant has measurable disease according to RECIST v1.1.
* Participant has documented radiographic evidence of disease progression from prior line of therapy.
* A biopsy (excisional, incisional, or core) of non-target tumor tissue obtained within 28 days prior to initiating lymphodepleting chemotherapy is mandatory if clinically feasible. This biopsy will be used as baseline for biomarker analyses. If it is not feasible to obtain a fresh biopsy, an archival tumor tissue (FFPE block) taken preferably after completion of the participant's last line of therapy, preferably within 90 days prior to initiating lymphodepleting chemotherapy, may be accepted.
* A haematologist has been consulted prior to lymphodepletion in participants who have had a serious/significant bleeding/thrombosis history.

Exclusion Criteria:

* Central nervous system (CNS) metastases.
* Any other prior malignancy that is not in complete remission.
* Previous treatment with genetically engineered NY-ESO-1-specific T cells.
* Previous NY-ESO-1 vaccine or NY-ESO-1 targeting antibody.
* Prior gene therapy using an integrating vector
* Previous allogeneic hematopoietic stem cell transplant
* Clinically significant systemic illness (serious active infections or significant cardiac, pulmonary, hepatic, or other organ dysfunction, that in the judgment of the Investigator would compromise the participant's ability to tolerate protocol therapy or significantly increase the risk of complications) or prior or active demyelinating disease
* Participant has received cytotoxic therapy within 3 weeks prior to lymphodepleting chemotherapy
* Systemic corticosteroids or any other immunosuppressive therapy within 2 weeks prior to lymphodepleting chemotherapy.
* Participant has received ≥50 Gy to a significant volume of the pelvis, long bones or spine, or a cumulative dose of radiation that, in the Investigator's opinion would predispose patients to prolonged cytopenia after lymphodepletion.
* All of the participant's measurable lesions have been irradiated within 3 months prior to lymphodepletion. An irradiated measurable lesion with unequivocal progression following irradiation may be considered a target lesion regardless of time from last radiotherapy dose.
* Participant has received an anti-cancer vaccine within 2 months in the absence of tumor response. The participant should be excluded if their disease is responding to an experimental vaccine given within 6 months.
* Participant has received live vaccine within 4 weeks prior to lymphodepletion or intends to receive live vaccine during the 3-month period following administration of lete-cel.
* Participant has received immune therapy (monoclonal antibody therapy, checkpoint inhibitors) within 4 weeks of lymphodepletion.
* Participant had major surgery ≥28 days of first dose of study intervention

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2019-12-31 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
ORR (Overall Response Rate) | Up to approximately 36 months
  ORR is defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) via investigator assessment per Response Evaluation Criteria in Solid Tumors Criteria (RECIST) version 1.1 relative to the total number of participants in the analysis population. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g., percent change from baseline). 95% CI is based on Clopper-Pearson exact confidence interval.

SECONDARY OUTCOMES:
DCR (Disease Control Rate) | Up to approximately 36 months
  DCR, is defined as the percentage of participants with a confirmed CR, PR, or SD with minimal 12 weeks duration relative to the total number of participants within the analysis population at the time of primary analysis as determined by independent central review per RECIST v1.1. The observed DCR will be reported along with 95% Clopper-Pearson exact confidence interval (CI). DCR will be analyzed based on PEAP and mITT populations.
PFS (Progression Free Survival) | Up to approximately 54 months
  PFS, is defined as the time from the date of T-cell infusion until the earliest date of radiological PD as assessed by independent central review per RECIST v1.1, or death due to any cause. For the analysis of PFS, if the participant received subsequent anticancer therapy prior to the date of documented events, PFS will be censored at the last adequate disease assessment (e.g., assessment when visit level response was CR, PR, or SD) prior to the initiation of the new anticancer therapy. If a participant does not have an adequate post-baseline disease assessment that is no later than the date of initiation of anti-cancer therapy, PFS will be censored at the date of the T-cell infusion date.
OS (Overall survival) | up to 15 years post-T-cell infusion
  OS is defined as the interval of time between the date of T-cell infusion and the date of death due to any cause. For participants who do not die, time of death will be censored at the date of last contact. The date of death should be taken from that recorded on the Record of Death page. Death on study due to any cause will be included. Survival will be listed and summarized using Kaplan-Meier quartile estimates along with 2-sided 95% CI.
DOR (Duration of response) | Up to approximately 54 months
  DOR is defined as, in the subset of participants who show a confirmed CR or PR as assessed by independent central review per RECIST v1.1, the time from first documented evidence of CR or PR until the first documented sign of disease progression or death. Duration of response will be summarized descriptively, if data warrant, using Kaplan-Meier medians and quartiles. Censoring: same as PFS censorship table.
TTR (Time to response) | Up to approximately 54 months
  TTR is defined as the time from the date of T-cell infusion to initial date of confirmed response (PR or CR) as assessed by independent central review per RECIST v1.1 in the subset of participants who achieved a confirmed PR or CR.
  TTR will be listed and summarized descriptively using median and quartiles in the subset of participants with a confirmed response of PR or CR.
  Efficacy listings such as BOR, DOR, PFS and OS will be reported for the PEAP and mITT populations.
Number of Participants with Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | Up to approximately 54 months
  An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations which involve medical or scientific judgment or is associated with liver injury and impaired liver function.
Number of Participants with AEs of Special Interest (AESIs) | Up to approximately 54 months
  An AESI may be of scientific and medical concern related to the treatment, monitored, and rapidly communicated by investigator to sponsor. AESIs included cytokine release syndrome (CRS), hematopoietic cytopenias (including pancytopenia and aplastic anemia), graft vs host disease (GVHD), ICANS, Guillain-Barre syndrome, treatment-related inflammatory response at tumor site(s), and neutropenia Grade 4 lasting ≥28 days.
Number of Participants with TEAEs and TESAEs by Severity | Up to approximately 54 months
  An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations which involve medical or scientific judgment or is associated with liver injury and impaired liver function. AEs and SAEs were graded according to National Cancer Institute-Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version 5.0. Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe or medically significant but not immediately life-threatening; Grade 4- Life-threatening consequences; Grade 5- Death related to AE.
Number of Participants with AESIs by Severity | Up to approximately 54 months
  An AESI may be of scientific and medical concern related to the treatment, monitored, and rapidly communicated by investigator to sponsor. AESIs included cytokine release syndrome (CRS), hematopoietic cytopenias (including pancytopenia and aplastic anemia), graft vs host disease (GVHD), ICANS, Guillain-Barre syndrome, treatment-related inflammatory response at tumor site(s), and neutropenia Grade 4 lasting ≥28 days.
Percentage of Participants with Replication Competent Lentivirus (RCL) Positive | Up to approximately 54 months
  RCL was monitored using a polymerase chain reaction (PCR)-based assay that detects and measures copies of the gene coding for the vector's envelope protein, namely vesicular stomatitis virus G protein (VSV-G).
Instances of Insertional Oncogenesis (IO) | Up to approximately 54 months
  Instances of Insertional Oncogenesis (IO) was summarized descriptively
Maximum Transgene Expansion (Cmax) | Day 1 to Day 14
  Cmax was defined as maximum observed persistence, determined directly from the persistence-time data. Blood samples were collected for PK analysis
Time to Cmax (Tmax) | Day 1 to Day 14
  Tmax was defined as time to reach Cmax, determined directly from the persistence-time data. Blood samples were collected for PK analysis.
Area Under the Time Curve from Zero to Time 28 Days (AUC [0-28]) | Up to 28 days
  Area under the persistence-time curve from time zero to Day 28. Blood samples were collected for PK analysis.

CONTACTS AND LOCATIONS:
Locations (38):
- United States (24):
  - City of Hope National Medical Center, Duarte, California
  - Stanford Hospital and Clinics, Stanford, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - University of Iowa College of Medicine, Iowa City, Iowa
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering cancer center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University-Columbus, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh, Hillman Cancer centre, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University Of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Froedtert Hospital, Milwaukee, Wisconsin
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - CIUSSS de L'Est-De-Lile-De-Montreal, Montreal, Quebec
- France (2):
  - Centre Léon Bérard, Lyon
  - CHU de Bordeaux GH Sud Hôpital Haut Lévêque, Pessac
- Italy (2):
  - Fondazione IRCCS Instituto Nazionale Dei Tumori, Milan, Lombardy
  - Ircss Istituto Clinico Humanitas, Rozzano (MI), Lombardy
- The Netherlands Cancer Institute, Amsterdam, Netherlands
- Spain (4):
  - Hospital Santa Creu Y Sant Pau, Barcelona
  - Ico Duran y Reynals l'Hospitalet de Llobrega, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Virgen Del Rocio, Seville
- United Kingdom (3):
  - Royal Marsden Hospital, London
  - University College Hospital-London, London
  - Christie Hospital NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No